CLINICAL TRIAL: NCT02480426
Title: Guidance for TIPS Creation: CT-image Versus CO2 Portography
Brief Title: 3D CT Guidance for Transjugular Intrahepatic Portosystemic Shunt Creation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-overlay
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT-image guidance (Experimental): Previously acquired portal venous phase of CT datasets and intra-operative CT datasets were registered on a dedicated workstation. The selected volume of interest of the CT-image showing portal vein vasculature was overlaid onto the fluoroscopic display as real-time 3D CT-image guidance during the procedure.
  Interventions: Device: CT-image guidance
- CO2 portography (Active Comparator): two two-dimensional (2D) CO2 portograms
  Interventions: Drug: CO2 portograms guidance

INTERVENTIONS:
Device: CT-image guidance — TIPS creation is performed under the guidance of 3D CT-image.
  Arms: CT-image guidance
Drug: CO2 portograms guidance — TIPS creation is performed under the guidance of two-dimensional (2D) CO2 portograms.
  Arms: CO2 portography

SUMMARY:
To prospectively evaluate the efficacy of real-time 3D CT-image guidance and CO2 portography during transjugular intrahepatic portosystemic shunt (TIPS) creation.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis
2. Scheduled for indicated TIPS procedure

Exclusion Criteria:

1. Presence of portal vein thrombosis
2. Presence of ascites
3. Presence of hepatic vein occlusion or stenosis
4. Proven malignancy including hepatocellular carcinoma 5. End-stage renal disease under renal replacement therapy; 6. Cardiorespiratory failure 7. Pregnancy or patients not giving informed consent for TIPS procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | procedure

SECONDARY OUTCOMES:
Median needle passes for portal vein entry | procedure
Median radiographic fluoroscopy time for portal vein entry | procedure
The median radiation dose for the whole TIPS procedure | procedure
The rate of TIPS complication | 6 months